CLINICAL TRIAL: NCT05095792
Title: Evaluation of the Effect of Ketamine on Neurological Activity as Measured by Quantitative EEG
Brief Title: Effect of Ketamine on Neurological Activity as Measured by Electroencephalogram (EEG)
Status: Terminated | Type: Observational
Why Stopped: Business decision to stop enrollment after 1 participant completed the study. Will not be reopening.
Sponsor: Entheon Biomedical Corp. (Industry)
Responsible Party: Sponsor
Other Study IDs: EBIQ-101
Record Dates: First submitted 2021-10-05; First posted 2021-10-27 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-11

CONDITIONS: Treatment-resistant Depression
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Observational - no intervention — This is an observational study with no intervention.

SUMMARY:
This observational study will allow data to be collected to demonstrate changes in brain activity following administration of standard of care (SOC) Ketamine. By comparing genetic markers across participants, data on impact of genetic markers and response to Ketamine will also be analysed. This data will contribute to the design of future studies utilizing Ketamine for various psychiatric disorders. This study will focus on treatment-resistant Major Depressive Disorder (MDD).

DETAILED DESCRIPTION:
This is an Open Label Observational Study with the primary objective to assess brain activity in patients prior to, during and after Ketamine treatment and to assess genetic markers prior to Ketamine treatment. This is a non-interventional study that will observe the Electroencephalogram (EEG) pattern of participants who, per standard of care, are treated with intramuscular Ketamine. The administration of the Ketamine during this study is not considered investigational. The experimental intervention, measurements via EEG, will be offered to patients of the study site presenting for intramuscular (IM) ketamine treatment per the site's established and evidence-based protocol as part of their regular clinical care. Participants in this study have already been determined to have a medically appropriate indication for IM Ketamine treatment, independent of enrollment in this study. Given the requirement, per study protocol, to wear an EEG headset and complete study measures, participants will be compensated by having treatment costs paid by the study sponsor. There will be 36 participants enrolled at one study site.

ELIGIBILITY:
Inclusion Criteria:

1. Primary Diagnostic and Statistical Manuel of Mental Disorders 5 (DSM-V) diagnosis of treatment-resistant Major Depressive Disorder (may have secondary diagnoses of general anxiety, substance disorder)

   * Non-responders to at least 2 previous anti-depressant medications prescribed by a physician in the past five years
   * Score of ≥20 on Montgomery-Asberg Depression Rating Scale (MADRS) (i.e., moderate to severe depression)
2. All genders aged 21 to 60 years of age
3. Prescribed Ketamine or currently being treated with Ketamine for treatment-resistant Major Depressive Disorder
4. Willing to wear an Electroencephalogram (EEG) headset and an eye mask
5. Willing to listen to ambient sound
6. Willing to have a genetic cheek swab

Exclusion Criteria:

1. Pregnancy
2. Traumatic Brain Injury within past 3 months
3. Body weight < 50 kg or > 120 kg
4. Coronary heart disease
5. Uncontrolled hypertension as defined in the American College of Cardiology/American Heart Association (ACC/AHA) Hypertension Guidelines
6. Previous contact with Ketamine (therapeutically or recreationally) outside of treatment at the study site
7. Primary psychotic disorder (e.g., schizophrenia, schizoaffective disorder)
8. Bipolar disorder with current manic, hypomanic or mixed state
9. Post-traumatic stress disorder
10. Obsessive-compulsive disorder
11. Primary substance-use disorder
12. Alcohol consumption 24 hours prior and 48 hours subsequent to treatment
13. Currently using any of the following medications:

    * Benzodiazepines for 6 hours prior to treatment and 2 hours after treatment
    * Lamotrigine for 6 hours prior to treatment
    * Amphetamine-based stimulants for 6 hours prior to treatment
    * Monoamine Oxidase Inhibitors (MAO-Is) may be taken but blood pressure must be monitored

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Male or female participants with treatment-resistant Major Depressive Disorder aged 21-60 interested in receiving intra-muscular injections of ketamine over 10 sessions in the clinic and willing to wear an electroencephalogram (EEG) headset to measure their brain wave patterns.
Sampling Method: Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2021-11-09 (Actual); Primary Completion 2022-10-21 (Actual); Study Completion 2022-10-21 (Actual)

PRIMARY OUTCOMES:
Inter and intra patient variability in neurological activity. | Up to 74 days
  Observation of the the inter and intra patient variability in neurological activity.

SECONDARY OUTCOMES:
Genetic markers on neurological phenotypes | Baseline
  Correlation of neurological phenotypes with genetic markers
CADSS-6 correlation with neurological phenotypes | Up to 67 days
  Correlation of neurological phenotypes of Clinician Administered Dissociative Symptom Scale (CADSS-6).
QIDS SR-16 correlation with neurological phenotypes | Up to 67 days
  Correlation of neurological phenotypes of depressed patients with Quick Inventory of Depressive Symptomatology (QIDS SR-16)
PMQ-SF correlation with neurological phenotypes | Up to 67 days
  Correlation of neurological phenotypes Psychedelic Music Questionnaire Short Form (PMQ-SF)

CONTACTS AND LOCATIONS:
Overall Officials: Steven Levine, MD, Principal Investigator — Heading Health
Locations (1):
- Heading Health, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-10-13): https://cdn.clinicaltrials.gov/large-docs/92/NCT05095792/Prot_SAP_000.pdf